CLINICAL TRIAL: NCT07198555
Title: A Clinical Study to Evaluate the Safety, Tolerability and Efficacy of BBM-A101 in the Treatment of Knee Osteoarthritis .
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability and Efficacy of BBM-A101 in the Treatment of Knee Osteoarthritis.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Belief BioMed (Beijing) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BBM007-CLN1001
Record Dates: First submitted 2025-09-19; First posted 2025-09-30 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; gene therapy; Adeno-Associated Virus
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Masking Description: The masking subjects in the Ia phase is participant , but the phase Ib study is double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm of Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm of BBM-A101 (Experimental)
  Interventions: Drug: BBM-A101

INTERVENTIONS:
Drug: BBM-A101 — Single-dose intra-articular （IA）injection （2ml）(phase Ia)
  Low dose group， Middle dose group； High dose group； Control group ：Placebo
  Arms: Arm of BBM-A101
Drug: Placebo — Placebo(phase Ia)
  Arms: Arm of Placebo
Drug: BBM-A101 — Single-dose intra-articular （IA）injection （2ml）(phase Ib) Low dose group， High dose group
  Control group ：Placebo
  Arms: Arm of BBM-A101
Drug: Placebo — Placebo（phase Ib）
  Arms: Arm of Placebo

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and efficacy of BBM-A101 to treat participants with knee osteoarthritis.

DETAILED DESCRIPTION:
This study is divided into two phases: Phase Ia and Phase Ib . Phase Ia is a randomized, single-blind study . Phase Ib is a randomized, double blind, parallel assignment study.

BBM-A101 is an AAVbased gene therapy that delivers a therapeutic gene cassette into knee for the treatment of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with moderate knee osteoarthritis .
2. The knee joint was evaluated as having Kellgren-Lawrence grade 2 or 3.
3. The Body Mass Index (BMI) ranges from 18.0 to 35.0 kg/m2 (including the boundary values).
4. Lower titers of antibodies binding to the BBM-A101 capsid in the blood.
5. Participants who had received adequate treatment with conventional medications previously, experienced recurrence or aggravation of target knee arthritis after discontinuation of medication, and still had moderate pain; during the screening period, the WOMAC pain score of the target knee was ≥ 8 .
6. From the time of screening to 52 weeks after dosing , the participants had no intention of having children and voluntarily took effective contraceptive measures, and there were no plans for sperm donation or ova donation.
7. Voluntarily sign the informed consent form and be able to complete the research as required by the clinical trial protocol.

   -

Exclusion Criteria:

1. There is a possibility of secondary knee osteoarthritis, or the knee joint symptoms may not be caused by knee osteoarthritis, or there may be other medical histories of diseases that other researchers believe could potentially lead to knee osteoarthritic inflammation.
2. History of lumbar dischernaiation, accompanied by lower limb nerve symptoms that may affect the assessment of the study.
3. Participants who are unable or unwilling to undergo MRI examination, or who have contraindications to MRI.
4. Participants who are unable or unwilling to undergo joint fluid extraction.
5. During the screening period and before dosing, there were clinically significant abnormal values in the laboratory tests, and the researchers believed that these might pose risks to the participants in the clinical trial.
6. Those with positive results for hepatitis B virus surface antigen or hepatitis B virus deoxyribonucleic acid or hepatitis C virus ribonucleic acid test or human immunodeficiency virus antibody or Treponema pallidum antibody.
7. Currently undergoing treatment for hepatitis B and hepatitis C.
8. Participants who had persistent chronic or active infections within the previous 4 weeks were selected.
9. Participants who had coagulation disorders (such as hemophilia) or existing medical conditions that require anticoagulation therapy and make knee joint injection impossible.
10. Having or having had cancer or malignant tumors
11. Having received genetic therapy or stem cell therapy before screening or having plans for genetic therapy or stem cell therapy during the study period.
12. Any history of vaccination within 30 days prior to dosing or any vaccination schedule within 30 days after dosing.
13. Screening will be conducted on female participants who are pregnant or breastfeeding or whose HCG test result is positive; or who have plans to get pregnant within the next 52 w.
14. History of alcohol addiction or drug dependence, or inability to limit alcohol consumption during the research process.
15. Participants had any mental disorders that might affect the assessment of the study.
16. Having other conditions that the investigator consider unsuitable for participation in the study.

    -

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) events | within 4 weeks
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | within 52 weeks
  To evaluate the safety of BBM-A101 by AEs and SAEs.

SECONDARY OUTCOMES:
The protein levels of gene expression products in blood and joint fluid | within5 years
The shedding of recombinant adeno-associated virus (rAAV) vectors in peripheral blood, joint fluid, urine, feces, saliva, and semen | within 5 years
The change in the joint space width as detected by X-ray of the knee joint compared to the baseline | within 5 years
The changes in the titers of AAV capsid-binding antibodies in the blood and joint fluid compared to the baseline level | within 5 years
The changes in the titers of antibodies binding to the expressed products in the blood and joint fluid compared to the baseline level | within 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jie Zhao, Principal Investigator — The Ninth People's Hospital of Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The Ninth People's Hospital of Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No